CLINICAL TRIAL: NCT00495755
Title: An Open Label Phase I Trial of Alemtuzumab (Campath 1-H) Therapy for Refractory Chronic Graft-vs-Host Disease
Brief Title: Campath in Chronic GVHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFCI 07-057
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Graft-vs.-Host Disease
Keywords: Chronic Graft-vs-Host Disease
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath (alemtuzumab) (Experimental)
  Interventions: Drug: Alemtuzumab (Campath)

INTERVENTIONS:
Drug: Alemtuzumab (Campath) — An escalating dose given over 4 weeks

SUMMARY:
The CD52 antigen, which is targeted by alemtuzumab, is highly expressed on mature T lymphocytes, monocytes and monocyte-derived dendritic cells as well as on mature B cells. Due to its more promiscuous effect on immune cells, alemtuzumab not only targets antibody producing B lymphocytes as does rituximab, but also targets alloreactive T lymphocytes and dendritic cells that also contribute to the complex pathogenesis of chronic GVHD.

Our hypothesis is that alemtuzumab will be effective in the treatment of chronic GVHD through its promiscuous depletion of alloreactive T lymphocytes, dendritic cells as well as antibody producing mature B-lymphocytes.

DETAILED DESCRIPTION:
This is a phase I, dose escalation trial of alemtuzumab for patients with steroid-refractory chronic GVHD. Alemtuzumab will be given over a 4-week period.

Three escalating doses of alemtuzumab will be considered to determine the maximum tolerated dose (MTD). In this design, a cohort of 3-6 patients will be treated at each dose level. Dose-limiting toxicity (DLT) will be defined as any life-threatening anaphylaxis due to an alemtuzumab infusion, any grade 4 non-hematologic toxicity directly related to alemtuzumab during the 12 week assessment period, any grade 4 hematological toxicity, and any grade 4 infectious complication that requires hospitalization. CMV reactivation secondary to alemtuzumab is an expected complication of alemtuzumab and will not be considered a DLT unless grade 4 CMV disease occurs. CMV DNA levels will be closely monitored and preemptive therapy for CMV will be initiated if there is evidence of CMV reactivation.

Three patients will be entered at each dose level. The dose of alemtuzumab will be escalated if these 3 patients complete the 4-week treatment and none experience a DLT by week 12 of therapy. If 1 of 3 patients treated at a given dose level experiences a DLT, then 3 more patients are treated at that dose level. If the incidence of DLT among those 6 patients is 1 in 6, then dose escalation to the next highest dose level occurs. If 2 or more of the 6 patients treated at a dose level experience DLT, then the MTD is considered to have been exceeded. At that point, unless 6 patients were treated at the previous dose level, 3 further patients will be treated at that level, and the same principles for determination of the MTD apply. There will be no further dose escalation at this point, and the MTD will be the dose level at which no more than 1/6 subjects experience a DLT. Once 6 patients have been treated at the MTD, an additional 10 patients will be treated at that dose level to further delineate toxicity and efficacy at that dose level.

Patients who experience either no toxicity, grade I-II toxicity that has resolved by the time of clinical response assessment and who have had no response or only a partial response to therapy can receive a second course of alemtuzumab after week 12. The second course of alemtuzumab will be a 4-week course at the same dose and schedule as the first course of treatment. Patients who have complete response and resolution of their chronic GVHD will not be retreated regardless of toxicity. Patients with any grade IV toxicity will not be retreated regardless of their response. Toxicity associated with second courses of therapy will not be used in the assessment of the MTD.

Toxicity assessments will be ongoing and recorded at scheduled clinical visits. Clinical response assessments will be done by assessing the presence or absence of signs and symptoms of GVHD after completion of 3 months on the study, during week 12. A similar series of immunologic assays will be performed on subjects enrolled on this clinical trial as in Specific Aim 1.

Eligible patients will have undergone allogeneic stem cell transplantation using myeloablative or non-myeloablative conditioning regimens at least 180 days (6 months) ago. Patients must have steroid refractory chronic GVHD, defined as having persistent signs and symptoms of chronic GVHD despite the use of prednisone at >0.5 mg/kg/day or 1 mg/kg every other day for at least 4 weeks in the preceding 12 months (or equivalent dosing of alternate corticosteroids) without complete resolution of signs and symptoms. Patients with either extensive chronic GVHD or limited chronic GVHD requiring systemic therapy are eligible. Subjects must be on stable doses of immunosuppressants and corticosteroids for 4 weeks prior to enrollment, and the dose of corticosteroids must be less than 2mg/kg/day prednisone use (or equivalent). Subjects will be required to have adequate bone marrow and organ function at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic stem cell transplantation using myeloablative or non-myeloablative conditioning regimens.
* Patients must be at least 180 days (6 months) from the allogeneic stem cell transplantation procedure.
* Patients must have steroid refractory chronic GVHD, defined as having persistent signs and symptoms of chronic GVHD despite the use of prednisone at < 0.5 mg/kg/day or 1 mg/kg every other day for at least 4 weeks in the preceding 12 months (or equivalent dosing of alternate corticosteroids) without complete resolution of signs and symptoms. Patients with either extensive chronic GVHD or limited chronic GVHD requiring systemic therapy are eligible.
* Stable dose of corticosteroids for 4 weeks prior to enrollment.
* Less than 2mg/kg/day prednisone use (or equivalent).
* No addition or subtraction of other immunosuppressive medications (e.g. calcineurin inhibitors, sirolimus, mycophenolate mofetil) for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug.
* Adequate bone marrow function indicated by:
* ANC>1000/mm3
* Platelets>50,000/mm3
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment

Exclusion Criteria:

* Prednisone requirement>2mg/kg/day or equivalent
* Known life-threatening hypersensitivity to alemtuzumab, other anti-B cell or anti-T cell antibodies.
* Prior exposure to any new immunosuppressive medication (or Extra Corporeal Phototherapy) in the preceding 4 weeks prior to enrollment.
* Active, uncontrolled infection.
* History of Hepatitis B or C infection.
* Active malignant disease relapse.
* Donor lymphocyte infusion within the preceding 100 days or plan for donor lymphocyte infusion in the coming 3 months.
* Life expectancy <3 months.
* Pregnancy or lactation.
* Evidence of HIV seropositivity.
* Inability to comply with alemtuzumab treatment regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-07; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD MPH FRCPC, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Campath (Alemtuzumab): 3 dose cohorts entered
Period: Overall Study
Arm/Group | Campath (Alemtuzumab)
Started | 13
Completed | 10
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Campath (Alemtuzumab)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of a Four-week Course of Alemtuxumab in Chronic GVHD for Patients With an Incomplete Response to Steroids
Description: MTD: The dose at which fewer or equal to 2/6 experience a dose-limiting toxicity
Time Frame: 12 weeks
Measure: Number; unit: mg
Arm/Group | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 13
mg | 53

2. Secondary Outcome: The Efficacy of a Four-week Course of Alemtuzumab in Patients With Steroid-refractory Chronic GVHD (cGVHD).
Description: Efficacy measured as complete response (CR), partial response (PR), stable disease (SD) and cGVHD progression (PD). CR is defined as absence of all measurable or symptomatic cGVHD, PR is defined as a remission in some but not all involved organs. SD is defined as no measurable change in GVHD and PD is defined as progression in at least one involved organ.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Response
Number analyzed (Participants) | 10
participants
  Complete Response | 3
  Partial Response | 4
  Stable Disease | 2
  cGVHD progression | 1

3. Secondary Outcome: The Effect of Alemtuzumab Therapy on Parameters of Cellular and Humoral Immunity in the Late Post Transplant Period. This Information is Exploratory in Nature Only Due to the Heterogeneity of the Anticipated Patient Population.
Time Frame: 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Campath (Alemtuzumab)
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath (Alemtuzumab) (N=13)
Parainfluenza (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Influenza A infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BK virus infection (Renal and urinary disorders) | 1 (1)
Adenovirus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pseudomonas infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
E.Coli bacteremia (Blood and lymphatic system disorders) | 1 (1)
Perirectal abscess (Gastrointestinal disorders) | 1 (1)
Corynebacterium infection (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes